CLINICAL TRIAL: NCT02801019
Title: Wear and Creep of Vitamin E-Diffused Highly Cross-Linked Polyethylene Liners Randomized Radiostereometric Study of 70 Hips Followed for 2 Years
Brief Title: Vitamin E-Diffused Highly Cross-Linked Polyethylene Liner
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sahlgrenska University Hospital (Other)
Responsible Party: Principal Investigator, Bita Shareghi, PhD student, Sahlgrenska University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: Dnr 279-08
Record Dates: First submitted 2014-04-30; First posted 2016-06-15 (Estimated); Last update posted 2016-06-15 (Estimated); Status verified 2016-06

CONDITIONS: Osteoarthritis
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- E-XLPE (Experimental): E-poly
  Interventions: Other: E-poly; Other: ArComXL
- C-XLPE (Active Comparator): ArComXL
  Interventions: Other: E-poly; Other: ArComXL

INTERVENTIONS:
Other: E-poly — comparison of two different polyethylene plastic 0,04 mm at 3 months 0,06 at 2 years
Other: ArComXL — comparison of two different polyethylene plastic 0,03 mm at 3 months 0,10 mm at 2 years

SUMMARY:
Vitamin E incorporated highly cross linked polyethylene (E-XLPE) was developed to increase oxidative resistance of highly cross-linked polyethylene (XLPE) without affecting mechanical properties. The investigators evaluated this type of polyethylene in a randomized clinical study, using Radiostereometric Analysis (RSA). The objective of this study was to compare the early-term wear of E-XLPE to a compression annealed polyethylene liner (C-XLPE, ArComXL®). The clinical outcome at two years was not expected to be affected by the choice of polyethylene.

DETAILED DESCRIPTION:
First generation of modern highly cross-linked polyethylene (XLPE) was clinically introduced in 1998 and has in most countries become standard as bearing surface in total hip arthroplasty. Studies of these materials have shown significantly reduced femoral head penetration when compared to gamma sterilized conventional polyethylene.

Thermaly treating (melting or annealing) is often a part of the manufacturing process of highly cross-linked polyethylenes. The polyethylene is exposed to irradiation to achieve cross-linking and improve wear resistance. Cross-linking by irradiation increases the amount of free radicals in the material.These radicals must be eliminated or stabilized to avoid oxidative degradation over time.Thermal treatment improves oxidation resistance but potentially changes the mechanical properties of the polyethylene.

By annealing i.e. heat treatment under the melt temperature the material maintains better mechanical properties, but elimination of free radicals is suboptimal, which can lead to oxidation in vivo.Heat treatment of the polyethylene above the melt temperature will more effectively reduce or eliminate the amount of residual free radicals. This will increase oxidation resistance, but will negatively influence the mechanical properties of the material.

Due to these limitations new generations of cross-linked polyethylene materials have been developed. Introducing Vitamin E (α-tocopherol), a natural antioxidant into the material prevents oxidative degradation and stabilizes the free radicals found in irradiated polyethylene plastic. In laboratory tests, polyethylene liners with incorporated vitamin-E have demonstrated similar wear, greater strength and better resistance to oxidation compared with the first generation cross-linked polyethylene. Currently, there are only laboratory studies on vitamin E diffused polyethylene available.

The hypothesis in this study is that the early-term E-XLPE wear is low and comparable to a heat-treated XLPE. The investigators also hypothesize that implant fixation and clinical outcome at two years will be unaffected by the choice of polyethylene.

The investigators therefore evaluated the early bedding in and wear in an uncemented arthroplasty supplied with liners made of vitamin E diffusion doped XLPE (E1®, Biomet, Warsaw, IN, USA). In the control group the investigators used the same uncemented hip prosthesis with polyethylene liners manufactured to achieve high levels of crosslinking without sacrificing the mechanical strength and extinguish residual free radicals (ArComXL® , Biomet, Warzaw, IN, USA).

ELIGIBILITY:
Inclusion Criteria:

* primary and certain subgroups of secondary osteoarthritis
* Patients aged 20-75 years

Exclusion Criteria:

* inflammatory arthritis
* cortisone or chemotherapy treatment
* known osteoporosis or osteomalacia

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2008-06; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Wear of vitamin E incorporated highly cross linked polyethylene | up to 2 years
  Evaluation of the early bedding in and wear in an uncemented arthroplasty supplied with liners made of vitamin E diffusion doped XLPE in comparsion to annealed polyethylene liner, ArComXL.

SECONDARY OUTCOMES:
Cup and stem translations | up to 2 years
  Evaluation of cup and stem translations of vitamin E incorporated highly cross linked polyethylene compared to annealed polyethylene liner ArComXL liner.

OTHER OUTCOMES:
Precision of the Radiostereometric analysis method | Postoperatively, whitin 3 to 5 days after surgery
  The differences between the postoperative double-examinations was used to compute the precision for the method.

CONTACTS AND LOCATIONS:
Overall Officials: Johan Kärrholm, Professor, Principal Investigator — Sahlgrenska University Hospital